CLINICAL TRIAL: NCT05118906
Title: A Double-blind, Placebo-controlled Pilot Trial of BP1.4979 for the Treatment of Binge Eating Disorder
Brief Title: Pilot Study on BP1.4979 Effect on Binge Eating Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P20-08 / BP1.4979; 2021-000472-11 (EudraCT Number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP1.4979 (Experimental): 15 mg BID active treatment
  Interventions: Drug: BP1.4979 active drug
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP1.4979 active drug — 2 tablets 15 mg of BP1.4979 per day
  Other Names: BP1.4979
  Arms: BP1.4979
Drug: Placebo — 2 tablets of placebo per day
  Arms: Placebo

SUMMARY:
This pilot study is to assess the efficacy and safety of BP1.4979 15 mg BID in female patients with moderate to severe binge eating disorder (BED), as defined according to DSM-5 guidelines.

DETAILED DESCRIPTION:
First clinical study to assess the effect of the BP1.4979 on BED in female patients over an 8 week-tretament period.

ELIGIBILITY:
Inclusion Criteria:

* Patient must voluntarily express a willingness to participate in this study, sign and date an informed consent prior to beginning any protocol required procedures.
* Female aged between 18 and 65 years, inclusive.
* Diagnosis of BED according to DSM-5 criteria
* BMI < 50 kg/m2.

Exclusion Criteria:

* Current diagnosis of bulimia nervosa or anorexia nervosa.
* History of bariatric surgery.
* Patient who is pregnant, lactating, or of childbearing potential who is not using adequate contraceptive measures. The following are considered adequate methods of birth control: 1. intrauterine device (IUD); 2. barrier protection; 3. contraceptive implantation system; 4. oral contraceptive pills; 5. surgically sterile patient; and 6. abstinence. All participants should have a negative pregnancy test prior to randomization
* Ongoing alcohol or tobacco addiction treatment (except Nicotine Replacement Therapy [NRT] with at least one-month stable dose prior to screening visit).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Binge Eating episodes per week | 8 weeks
  Number of Binge Eating episodes per week as measured during baseline and at the end of the treatment period

SECONDARY OUTCOMES:
Binge Eating days per week | 8 weeks
  Number of Binge Eating days per week as measured during baseline and at the end of the treatment period
Quality of Life improvement (CGI-I) | 8 weeks
  Quality of life as per assessment on the Clinical Global Improvement (CGI-I) scale measured at randomization and at the end of the treatment period. The CGI is a 7-point scale that requires the clinician to assessment of the patient's illness at the beginning of the intervention (Baseline state) and rated as: 1, Normal, not at all ill; 2, Borderline mentally ill; 3, Mildly ill; 4, Moderately ill; 5, Markedly ill; 6, Severely ill; 7, Among the most extremely ill patients.
  The Clinical Global Impression-Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

OTHER OUTCOMES:
Safety assessed by AEs collection | 8 weeks
  Safety of BP1.4979 based on AEs reporting during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Clément, MD, PhD, Principal Investigator — Nutrition Department, La Pitié Salpêtrière Hospital, Paris
Locations (1):
- Nutrition Department, La Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No